CLINICAL TRIAL: NCT07163702
Title: Efficacy and Safety of Xinglou Chengqi Granule for Acute Ischemic Stroke (EXACT): a Multi-center, Randomized, Double-blinded, Dose-exploration Ⅱa Trial
Brief Title: Efficacy and Safety of Xinglou Chengqi Granule for Acute Ischemic Stroke
Acronym: EXACT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ying Gao, Professor, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025DZMEC-251-02
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; Xinglou Chengqi granules; randomized controlled trial
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-dose group (Experimental): 16 g of Xinglou Chengqi granules will be given to participants in the high-dose group.
  Interventions: Drug: High-dose Xinglou Chengqi granules
- Low-dose group (Active Comparator): 8 g of Xinglou Chengqi granules and 8 g of placebo will be given to participants in the low-dose group.
  Interventions: Drug: Low-dose Xinglou Chengqi granules and placebo

INTERVENTIONS:
Drug: High-dose Xinglou Chengqi granules — Patients will receive orally high-dose Xinglou Chengqi granules, combined with guidelines-based standard care.
  Other Names: Guidelines-based standard care
  Arms: High-dose group
Drug: Low-dose Xinglou Chengqi granules and placebo — Patients will receive orally low-dose Xinglou Chengqi granules, combined with guidelines-based standard care.
  Other Names: Guidelines-based standard care
  Arms: Low-dose group

SUMMARY:
This is a Ⅱa clinical trial. The purpose of this study is to preliminarily explore the optimal dosage of Xinglou Chengqi Granules in the treatment of acute ischemic stroke and to evaluate the efficacy and safety of Xinglou Chengqi Granules for acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients diagnosed with acute ischemic stroke.
2. Meet the criteria of TCM phlegm-heat and fu-organ excess syndrome.
3. Acute ischemic stroke within 7 days after onset.
4. 6 ≤ NIHSS <20.
5. Aged 18-70 years, male or female.
6. The patient or representative has signed informed consent.

Exclusion Criteria:

1. Suspected secondary stroke caused by brain tumor, brain trauma, hemopathy, etc.
2. NIHSS Ⅰa ≥2.
3. Already dependent in activities of daily living before the present acute stroke (defined as modified Rankin Scare score ≥2 )
4. Received or planned thrombolysis or endovascular therapy after onset.
5. Known severe liver or kidney dysfunction (alanine aminotransferase or aspartate transaminase > 2.5 times the upper limit of normal value, serum creatinine > 1.5 times the upper limit of normal value)
6. With cancers or uncontrolled diabetes.
7. The expected survival time is less than 3 months.
8. Patients who have used other traditional Chinese medicine for treating acute ischemic stroke since stroke onset.
9. Patients with severe mental disorders, dementia, or other comorbid diseases that may affect neurological function examination.
10. With a history of alcohol or drug abuse or drug dependence.
11. Those known to be allergic to the investigated drug or its components.
12. Pregnancy, potential pregnancy, or breastfeeding.
13. Currently participating in other clinical trials during the past 3 months.
14. Those who are judged by researchers to have poor compliance or are not suitable for participating in this study for any other reason.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The change of NIHSS score from baseline to day 14. | Baseline and Day 14.
  The change of the National Institutes of Health stroke scale (NIHSS) score from baseline to day 14 will be analyzed between groups.

SECONDARY OUTCOMES:
The proportions of patients with mRS ≤ 2 or mRS ≤ 1. | Day 30, Day 60 and Day 90.
  The proportions of patients with modified Rankin Scale (mRS) ≤ 2 or mRS ≤ 1 will be analyzed between groups.
The change of NIHSS score | Day 7, day 30, day 60, day 90.
  The change of NIHSS score will be analyzed at days 7, 30, 60, and 90.
The proportion of patients with Barthel Index score ≥ 95 or ≥ 75. | day 7, day 14, day 30, day 60, day 90.
  The proportion of patients with Barthel Index score ≥ 95 or ≥ 75 will be analyzed at days 7, 14, 30, 60, and 90.
The change of EQ-5D score. | day 7, day 14, day 30, day 60, day 90.
  The change of EQ-5D score from baseline to days 7, 14, 30, 60, and 90 will be analyzed between groups.
The incidence of new cardiovascular events. | day 7, day 14, day 30, day 60, day 90.
  The incidence of new cardiovascular events will be analyzed at day 7, 14, 30, 60, and 90.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongzhimen Hospital, Beijing University of Chinese Medicine, Richmond, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided